CLINICAL TRIAL: NCT03828045
Title: Routine Clinical Practice in Spain: Evaluation of the Use of Apremilast in Patients With Psoriatic Arthritis, Naïve to Biological Treatment (PREVAIL Study)
Brief Title: A Study to Evaluate the Use of Apremilast in Patients With Psoriatic Arthritis, Naïve to Biological Treatment
Acronym: PREVAIL
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSA-015; U1111-1221-8638 (Registry Identifier: WHO)
Record Dates: First submitted 2018-10-24; First posted 2019-02-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic Arthritis; Apremilast; CC-10004; Biologic Treatments
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Psoriatic Arthritis patients on Apremilast: Patients diagnosed with PsA (according to the CASPAR diagnosis criteria), naïve to biological treatments, who have - following the routine practice in their centers - initiated treatment with apremilast 6 months (±1 months) before their inclusion in the study, irrespective of treatment duration.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast

SUMMARY:
Observational, prospective and multicenter study in approximately 25 sites nationwide. The investigators participating in this study will be rheumatologists specializing in this pathology.

The study will include patients diagnosed with PsA (according to the CASPAR diagnosis criteria), naïve to biological treatments, who have - following the routine practice in their centers - initiated treatment with apremilast 6 months (±1 months) before their inclusion in the study, irrespective of treatment duration.

Recruitment will be consecutive and the reason for not including a potential candidate patient will be registered. The decision to prescribe apremilast treatment should be clearly dissociated from the inclusion of the patient in the study, which will not occur earlier than 6 months (± 4 weeks after treatment start). Therefore, the choice of the therapeutic strategy will be made independently by the physician.

Before entering the study, all patients shall sign an informed consent to participate in the study, including permission to retrieve data from their medical records and to complete questionnaires regarding their quality of life.

To avoid recruitment biases and obtain a homogeneous cohort regarding treatment duration, all consecutive patients who attend to a routine follow-up visit and have been prescribed apremilast 6 months (+/- 4 weeks) before the baseline visit, will be offered to enter the study. All consecutive patients who can be contacted 6 months (+/- 4 weeks) following initiation of treatment with apremilast will be approached for entry to minimize bias in patient selection

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years.
* Patients diagnosed with psoriatic arthritis according to the CASPAR criteria*.
* Patients who, following the routine clinical practice, initiated treatment with apremilast 6 months (±4 weeks) before their inclusion in the study.
* Patients naive to biologic treatments.

Exclusion Criteria:

* Patients who reject to sign the informed consent.
* Patients enrolled in a clinical trial within the 4 weeks preceding the baseline visit or for the duration of apremilast treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational, prospective and multicenter study in approximately 25 sites nationwide. The investigators participating in this study will be rheumatologists specializing in this pathology.
  The study will include patients diagnosed with PsA (according to the CASPAR diagnosis criteria), naïve to biological treatments, who have - following the routine practice in their centers - initiated treatment with apremilast 6 months (±1 months) before their inclusion in the study, irrespective of treatment duration.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Treatment persistence at 6 months after initiating apremilast treatment | Up to approximately 6 months
  Percentage of patients still being treated with apremilast after 6 months of initiating treatment

SECONDARY OUTCOMES:
Demographic characteristics | Up to approximately 6 months
  Description of the demographic at time of initiating treatment with apremilast
To describe the characteristics of apremilast treatment (i.e., dosage and regimen) in patients with PsA who start treatment according to the routine clinical practice. | Up to approximately 12 months
  To capture the changes in dose and regimen of apremilast.
To assess the persistence of apremilast treatment after 12 months of treatment start | Up to approximately 12 months
  Percentage of patients still being treated with apremilast after 12 months of initiating treatment
To assess the disease activity at 6 and 12 months of treatment with apremilast. | At 6 and 12 months
  The disease activity will be assessed by the DAPSA scale when the information available in the patient's medical record allows the estimation of the DAPSA score. Otherwise, the individual items of the DAPSA scale will be described separately.
Changes on clinical enthesitis and dactilitis | UP to approximately 12 months
  Assessment of the changes on clinical enthesitis and dactilitis count after 6 and 12 months of treatment with apremilast.
Tender joints count | Up to approximately 12 months
  Change from baseline in the joints deemed tender as per joint count assessment by physical exam.
Swollen joints count | UP to approximately 12 months
  Change from baseline in the joints deemed tender as per joint count assessment by physical exam.
Changes in the plasma concentration of C-reactive protein. | Up to approximately 12 months
  Assessment of the change in the plasma concentration of C-reactive protein after 6 and 12 months of apremilast treatment.
Physician Global Assessment of Disease Activity (PGA). | Up to approximately 12 months
  Assessment of the Physician Global Assessment of Disease Activity (PGA) after 6 and 12 months of apremilast treatment.
To assess the presence of erosive changes after 6 and 12 months of treatment with apremilast. | UP to approximately 12 months
  Joint erosion will be assessed radiologically, as regularly assessed in the routine practice of each center.
The VITACORA-19 questionnaires | UP to approximately 12 months
  are used to assess the health-related quality of life of patients with PsA in the setting of clinical trials
The Psoriatic Arthritis Impact of Disease (PsAID)-9 questionnaires | UP to approximately 12 months
  was developed under a 13-country EULAR initiative to evaluate the impact of psoriatic arthritis in clinical practice . The version used in this study (PsAID-9) consists of 9 items addressing pain, fatigue, skin problems, work and/or leisure activities, functional capacity, discomfort, sleeping disturbances, coping, and anxiety
Assessment of changes on affected joints | Up to approximately 12 months
  Assessment of the changes on affected joints count after 6 and 12 months of treatment with apremilast.
Assessment of DAPSA/cDAPSA scores | Up to approximately 12 months
  Assessment of the changes of the DAPSA/cDAPSA score at 6/12 month after treatment.
To assess the relationship between the count of affected joints DAPSA/cDAPSA score after 6 and 12 months of treatment with apremilast. | Up to approximately 12 months
  Assessment of the relationship between the count of affected joints at treatment start and the DAPSA/cDAPSA score after 6 and 12 months of treatment with apremilast. The Pearson or Spearman correlation will be performed to evaluate the relationship between these variables
Adverse events (AEs) | Up to approximately 12 months
  Number participants with adverse events.
To assess the changes in patient's assessment of disease activity after 6 and 12 months of apremilast treatment. | UP to approximately 12 months
  To assess the changes in patient's assessment of disease activity after 6 and 12 months of apremilast treatment. Assessment of the relationship between the count of affected joints at treatment start and the DAPSA/cDAPSA score after 6 and 12 months of treatment with apremilast.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (20):
- Spain (20):
  - H Son Espases, Mallorca, Balearic Islands
  - H Son Llatzer, Mallorca, Balearic Islands
  - H Txagorritxu de Vitoria, Vitoria-Gasteiz, Basque Country
  - H Univ Canarias, Santa Cruz de Tenerife, Canary Islands
  - H Parc Tauli, Barcelona, Catalonia
  - H Bellvitge, L'Hospitalet Del Llobregat, Catalonia
  - H Santa Maria Lleida, Lleida, Catalonia
  - H Joan XXIII, Tarragona, Catalonia
  - H Mérida, Badajoz, Extremadura
  - H Virgen del Puerto, Cáceres, Extremadura
  - H Virgen de la Arrixaca, El Palmar, Murcia
  - H Navarra, Pamplona, Navarre
  - H Perpetuo Socorro, Badajoz
  - H Del Mar, Barcelona
  - H Donostia, Donostia / San Sebastian
  - H Can Misses, Ibiza Town
  - H Santa Lucía, Murcia
  - H Monte Naranco, Oviedo
  - H l Esperit Sant, Santa Coloma de Gramenet
  - Universitaire Vaudoise*, Vigo

REFERENCES:
- [Derived] Gratacos-Masmitja J, Beltran Catalan E, Alvarez Vega JL, Urruticoechea-Arana A, Fito C, Maceiras F, Belzunegui Otano JM, Fernandez Melon J, Chamizo Carmona E, Abad Hernandez MA, Ros Vilamajo I, Castro Oreiro S, Pascual Alfonso E, Torre Alonso JC; PREVAIL team. Real-world apremilast use in biologic-naive psoriatic arthritis patients. Data from Spanish clinical practice. Reumatol Clin (Engl Ed). 2024 Jan;20(1):24-31. doi: 10.1016/j.reumae.2023.09.004. PMID 38233009
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com